CLINICAL TRIAL: NCT03426774
Title: Non-Invasive Determination of Nitric Oxide Release by Simulated Passive Jogging & Jumping Devices
Brief Title: Simulated Passive Jogging & Jumping Devices & NO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sackner Wellness Products LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GJHP2017; 20170208 (Other: WIRB)
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity; Blood Pressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Evaluation of the effects of GentleJogger and Gentle Jumper on noninvasive biometric data in various postures in two specify age groups a) Younger 25-59 yrs b) Older > 60 yrs Each Subject will serve as his or her own Sham Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- YG ( 25-59yrs) -GJogger (Experimental): Gentle Jogger applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jogger
- OG (Greater than 60 yrs)-GJogger (Experimental): Gentle Jogger applied to each individual in (1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jogger
- YG ( 25-59yrs) -GJumper (Experimental): Gentle Jumper applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jumper
- OG (Greater than 60 yrs)-Gjumper (Experimental): Gentle Jumper applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jumper
- YG ( 25-59yrs) -GJogger Sham (Sham Comparator): A Sham Gentle Jogger is applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jogger
- OG (Greater than 60 yrs)- GJogger-Sham (Sham Comparator): A Sham Gentle Jogger is applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jogger
- YG ( 25-59yrs) -GJumper- Sham (Sham Comparator): A Sham Gentle Jumper is applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jumper
- OG (Greater than 60 yrs)-GJumper Sham (Sham Comparator): A Sham Gentle Jumper is applied to each individual in 1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg Each Subject serves as his/her own control.
  Interventions: Device: Gentle Jumper

INTERVENTIONS:
Device: Gentle Jogger — Passive Simulated Jogging device (Gentle Jogger)
  Arms: OG (Greater than 60 yrs)- GJogger-Sham; OG (Greater than 60 yrs)-GJogger; YG ( 25-59yrs) -GJogger; YG ( 25-59yrs) -GJogger Sham
Device: Gentle Jumper — Passive Simulated Jumping Device ( Gentle Jumper)
  Arms: OG (Greater than 60 yrs)-GJumper Sham; OG (Greater than 60 yrs)-Gjumper; YG ( 25-59yrs) -GJumper; YG ( 25-59yrs) -GJumper- Sham

SUMMARY:
Movement is important for overall health. Lack of movement has been shown to be associated with numerous diseases. This study will assess the validity and usefulness of two innovative low risk, non-invasive wellness devices, the Gentle Jogger® and the Gentle Jumper that passively simulate the physical activities of jogging and jumping, respectively. The study will evaluate whether or not each of the devices in different body postures (seated, lying down, slight recumbent and slight head down) produces changes in blood pressure, and indices of dilatation of blood vessels, in a younger (25-59yr) and older (> 60 yrs.) subject population. Volunteers will be paid for their participation in the study.

A substudy of this larger study ( Effects of Gentle Jogger on blood pressure), will determine the effects of 30 min of gentle jogger in seated and supine posture compared to Sham

DETAILED DESCRIPTION:
Physical inactivity is a significant risk for various cardiovascular diseases including hypertension, diabetes, and stroke. To address the sitting disease Sackner Wellness Products has patented 2 non-invasive methods for inducing passive movement while in seated or supine posture the Gentle Jogger® and Gentle Jumper®, each simulating the activities of jogging and jumping respectively. Passive simulation of jogging and jumping introduces pulses into the circulation as the feet strike a semi-rigid surface within the chassis of the device. These pulsations stimulate release of beneficial mediators which are important to cardiovascular health. The study will recruit healthy subjects in a younger age group (25-59 yrs ) and older age group (> 60 yrs) in order to measure changes in blood pressure, cardiovascular indices of vasodilation, heart rate variability, and other non-invasively acquired biometric information in different postures [(1) supine, 2) semi-recumbent, 3) sitting, 4) Trendelenburg and 5) reverse Trendelenburg )], while at rest and during and after use of the GJogger and GJumper. Additionally, a subgroup of subjects will be asked to perform texting of a specified script in order to determine whether or not GJogger is a distraction during text messaging.

Participants will also be recruited for a sub-study of the above larger study. This sub-study will determine the effects of a single device Gentle Jogger in setaed and supine posture over a 30 min period on continuously measured non-invasive blood pressure, and compared the latter to SHAM. On day 1 Subjects will be randomized to begin in seated or supine posture with 30 min of SHAM, and 30 min of Gentle Jogger, 3 days latter the subject will cross over to start with the opposite posture of day 1.

This study will determine the effects of 30 min of sedentary supine or seated (SHAM) and the effects of 30 min of G. Jogger in these two postures on continuous noninvasive measured blood pressure

Volunteers will be paid for their participation in the study The Gentle Jogger and Gentle Jumper are non-FDA regulated wellness devices (2016) in which, 1) GJogger and GJumper as part of a healthy lifestyle may help to prevent certain chronic diseases or conditions such as heart disease, high blood pressure, and type 2 diabetes and, 2) may help living well with certain chronic diseases or conditions such as s heart disease, high blood pressure, and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 25 yrs
* Able to provide Informed Consent

Exclusion Criteria:

* Age less than 25 yrs
* Not able to provide informed consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
a/b ratio from Photoplethysmogragh | 3 hr
  Determination of the change in a/b ratio from the non invasively acquired arterial pulse waveform

SECONDARY OUTCOMES:
Blood Pressure Changes | 3 hr
  Determination of the changes in non invasively acquired continous blood pressure during and after use of the device in various postures

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Adams, M.D., Principal Investigator — Sackner Wellness Products LLC
Locations (1):
- CIC Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Adams JA, Lopez JR, Nadkarni V, Zolkipli-Cunningham Z, Ischiropoulos H, Sackner MA. The effects of a motorized passive simulated jogging device on descent of the arterial pulse waveform dicrotic notch: A single arm placebo-controlled cross-over trial. Physiol Rep. 2022 Aug;10(15):e15418. doi: 10.14814/phy2.15418. PMID 35924333
- [Derived] Sackner MA, Patel S, Adams JA. Changes of blood pressure following initiation of physical inactivity and after external addition of pulses to circulation. Eur J Appl Physiol. 2019 Jan;119(1):201-211. doi: 10.1007/s00421-018-4016-7. Epub 2018 Oct 22. PMID 30350153